CLINICAL TRIAL: NCT06676215
Title: Efficacy of Amino Acid Supplementation on Gut Function and Nutritional Status in FIlipino Children Below Three Years Old
Brief Title: Amino Acid Supplementation in Children with Stunting
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Food and Nutrition Research Institute, Philippines (Other Government)
Collaborators: International Atomic Energy Agency (Other Government); University of Glasgow (Other); Ghana Atomic Energy Commission (Unknown); Kamuzu University of Health Sciences (Other); University of Zambia (Other); Rutgers, The State University of New Jersey (Other); St. John's Research Institute (Other); cnesten, Morocco (Unknown)
Responsible Party: Principal Investigator, Amster Fei Baquiran, Senior Science Research Specialist, Food and Nutrition Research Institute, Philippines
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIERC-2023-004
Record Dates: First submitted 2024-10-04; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Stunted Growth
Keywords: Amino Acid Supplementation; Gut Function; Nutritional Interventions; Stunting; Children Below 3 Years Old
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): complementary food supplemented with indispensable amino acid (IAA) mix
  Interventions: Dietary Supplement: IAA mix supplement; Other: Complementary food comprised of rice and legumes
- Control Group (Experimental): complementary food without IAA mix
  Interventions: Other: Complementary food comprised of rice and legumes

INTERVENTIONS:
Dietary Supplement: IAA mix supplement — The intervention is a daily IAA dose that provides x1.5 the estimated average requirement (EAR) for a healthy child. This IAA dose will be mixed to the complementary food and will be taken once daily for 4 weeks (28 days) by the child in the intervention group.
  Arms: Intervention Arm
Other: Complementary food comprised of rice and legumes — Each study child will receive standard complementary food which he/she will take once daily for 4 weeks (28 days)

SUMMARY:
The goal of this intervention study is to determine the effects of indispensable amino acid (IAA) supplementation on children of either sex, aged 18 to 36 months. The main questions it aims to answer are:

* Does IAA supplementation affect biomarkers of Environmental Enteric Dysfunction (EED), through the Dual Sugar Lactulose/Rhamnose (L/R) test, plasma intestinal fatty acid binding protein, plasma lipopolysaccharide binding protein, fecal myeloperoxidase, fecal neopterin, and gut microbiota?
* Does IAA supplementation impact amino acid digestion, as assessed by a dual-stable isotope tracer?
* What is the weight gain and the changes in length-for-Age z-scores (LAZ) and body composition?

The researchers will compare the effects of consumption of standard complementary food with added IAA against a control group that has no added IAA through the assessment of the various biomarkers.

Participants will:

* answer questions regarding personal, demographic, anthropometric, and food intake information.
* provide biological samples, including breath, urine, stool, blood, and saliva.
* consume solutions or meals that contain sugars and/or stable isotope tracers.
* visit the FNRI and receive house visits by study staff.
* consume complementary food with or without supplement daily for 28 days.

DETAILED DESCRIPTION:
Protocol treatment will start within two weeks of enrollment to the study. Following the baseline study assessments, each participant will receive the standard complementary foods (in the control group) or standard complementary foods supplemented with IAAs (histidine, isoleucine, leucine, lysine, methionine, phenylalanine, threonine, tryptophan, and valine) (in the intervention group).

Standard complementary foods will be comprised of ingredients mainly of rice and legumes. Standard complementary foods are foods that meet the dietary needs of children 6-36 months of age.

At least three observed (controlled) feeding sessions per week will be conducted over the 4 weeks of the study to confirm that the entire supplement was consumed or confirm intake. The observed feeding will take place at the child's home or at the barangay center. Uptake on non-observed days will be based on the caregiver's report. On each intervention monitoring day, a questionnaire will also be administered to assess child morbidity that day and on the day prior. A pediatrician or an alternate medical practitioner will also be invited during the data collection where in stable isotopes will be administered. The duties and responsibilities of the physician include: medical assessment of the participant, assistance in the collection of blood samples, assessment of adverse events (if any), and provision of first aid (if needed).

In the absence of treatment delays due to adverse events, the intervention will continue for 1 month or until one of the following criteria apply:

* Child is not able to tolerate the supplement (throws up)
* Severe acute malnutrition (SAM)
* Inter-current illness that prevents further administration of treatment
* Unacceptable adverse event(s)
* Study participant voluntarily withdraws from treatment OR
* Other general or specific changes in the study participant's condition render the study participant unacceptable for further treatment in the judgment of the investigator.

For each participant, tests to be conducted at study enrolment will be spread over three days. At the end of the study, endline tests will be spread over 2 days. Baseline visits for breath, blood, urine, and fecal collection should be conducted within -3 days prior to study treatment (day 3) while endline visits should be conducted within +7 days of study treatment (day 31). The intervention will be provided in coded sachets, distributed as per convenient for local custom to best ensure compliance with a minimum of three supervised feeds per week to ensure supplement is consumed at least periodically by the child and also to assess compliance.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 36 months old (of either sex)
* Stunted (LAZ of less than -2)
* Parent, caregiver or guardian able and willing to give written, informed consent

Exclusion Criteria:

* Wasted (WHZ of less than -2)
* Overweight (WHZ of more than 2)
* Have had diarrhea (by self-report) in the preceding month
* Sibling or twin of another participating study child (2 children of different families in the same household are both eligible)
* Have taken antibiotics in the preceding month
* Have food allergies/intolerance
* Had a serious illness within the last three (3) months or have any underlying condition which in the opinion of the pediatrician would put the subject at undue risk of failing study completion or would interfere with analysis of study results

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Gut Permeability as Assessed by the Lactulose/Rhamnose (L/R) Test at 28 days | Baseline and end of intervention at 28 days

SECONDARY OUTCOMES:
Change from Baseline in Protein Absorption as Assessed by the Dual Stable Isotope Tracer (DSIT) Technique at 28 days | Baseline and end of intervention at 28 days
Change from Baseline in Gut Digestive Capacity Measured by the 13C-Sucrose Breath Test (SBT) at 28 days | Baseline and end of intervention at 28 days
Change from Baseline in Gut Function Based on Plasma LPS-Binding Protein (LPSBP) Concentration at 28 days | Baseline and end of intervention at 28 days
Change from Baseline in Gut Function Based on Intestinal Fatty Acid Binding Protein (iFABP) Concentration at 28 days | Baseline and end of intervention at 28 days
Change from Baseline in Gut Inflammation Based on Fecal Myeloperoxidase Concentration at 28 days | Baseline and end of intervention at 28 days
Change from Baseline in Gut Inflammation Based on Fecal Neopterin Concentration at 28 days | Baseline and end of intervention at 28 days

OTHER OUTCOMES:
Change from Baseline in Length-for-age z-score (LAZ) at 28 Days and 6 Months | Baseline and end of intervention at 28 days and follow-up after 6 months
Change from Baseline in Weight at 28 days | Baseline and end of intervention at 28 days
Change from Baseline in Body Composition in 6 months | Baseline and follow-up after 6 months
Correlation Between Gut Microbiota Composition and Plasma Biomarkers of Gut Function (LPSBP and iFABP) | Baseline, pre-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Amster Fei P. Baquiran, BS Chemistry, Principal Investigator — Department of Science and Technology Food and Nutrition Research Institute
Locations (1):
- Department of Science and Technology - Food and Nutrition Research Institute, City of Taguig, National Capital Region, Philippines

REFERENCES:
- [Background] Abtahi S, Sailer A, Roland JT, Haest X, Chanez-Paredes SD, Ahmad K, Sadiq K, Iqbal NT, Ali SA, Turner JR. Intestinal Epithelial Digestive, Transport, and Barrier Protein Expression Is Increased in Environmental Enteric Dysfunction. Lab Invest. 2023 Apr;103(4):100036. doi: 10.1016/j.labinv.2022.100036. Epub 2023 Jan 10. PMID 36870290
- [Background] Antiporta DA, Ambikapathi R, Bose A, Maciel B, Mahopo TC, Patil C, Turab A, Olortegui MP, Islam M, Bauck A, McCormick B, Caulfield LE; MAL-ED Network Investigators. Micronutrient intake and the probability of nutrient adequacy among children 9-24 months of age: results from the MAL-ED birth cohort study. Public Health Nutr. 2021 Jun;24(9):2592-2602. doi: 10.1017/S1368980020000877. Epub 2020 Jul 2. PMID 32611463
- [Background] Arnold BF, Null C, Luby SP, Unicomb L, Stewart CP, Dewey KG, Ahmed T, Ashraf S, Christensen G, Clasen T, Dentz HN, Fernald LC, Haque R, Hubbard AE, Kariger P, Leontsini E, Lin A, Njenga SM, Pickering AJ, Ram PK, Tofail F, Winch PJ, Colford JM Jr. Cluster-randomised controlled trials of individual and combined water, sanitation, hygiene and nutritional interventions in rural Bangladesh and Kenya: the WASH Benefits study design and rationale. BMJ Open. 2013 Aug 30;3(8):e003476. doi: 10.1136/bmjopen-2013-003476. PMID 23996605
- [Background] Arsenault JE, Brown KH. Effects of protein or amino-acid supplementation on the physical growth of young children in low-income countries. Nutr Rev. 2017 Sep 1;75(9):699-717. doi: 10.1093/nutrit/nux027. PMID 28938793
- [Background] Budge S, Parker AH, Hutchings PT, Garbutt C. Environmental enteric dysfunction and child stunting. Nutr Rev. 2019 Apr 1;77(4):240-253. doi: 10.1093/nutrit/nuy068. PMID 30753710
- [Background] Capanzana MV, Aguila DV, Gironella GMP, Montecillo KV. Nutritional status of children ages 0-5 and 5-10 years old in households headed by fisherfolks in the Philippines. Arch Public Health. 2018 Apr 16;76:24. doi: 10.1186/s13690-018-0267-3. eCollection 2018. PMID 29686867
- [Background] Denno DM, VanBuskirk K, Nelson ZC, Musser CA, Hay Burgess DC, Tarr PI. Use of the lactulose to mannitol ratio to evaluate childhood environmental enteric dysfunction: a systematic review. Clin Infect Dis. 2014 Nov 1;59 Suppl 4:S213-9. doi: 10.1093/cid/ciu541. PMID 25305289
- [Background] Devi S, Varkey A, Sheshshayee MS, Preston T, Kurpad AV. Measurement of protein digestibility in humans by a dual-tracer method. Am J Clin Nutr. 2018 Jun 1;107(6):984-991. doi: 10.1093/ajcn/nqy062. PMID 29771297
- [Background] Dewey KG, Brown KH. Update on technical issues concerning complementary feeding of young children in developing countries and implications for intervention programs. Food Nutr Bull. 2003 Mar;24(1):5-28. doi: 10.1177/156482650302400102. PMID 12664525
- [Background] Elango R. Tolerable Upper Intake Level for Individual Amino Acids in Humans: A Narrative Review of Recent Clinical Studies. Adv Nutr. 2023 Jul;14(4):885-894. doi: 10.1016/j.advnut.2023.04.004. Epub 2023 Apr 14. PMID 37062432
- [Background] Fahim SM, Das S, Sanin KI, Gazi MA, Mahfuz M, Islam MM, Ahmed T. Association of Fecal Markers of Environmental Enteric Dysfunction with Zinc and Iron Status among Children at First Two Years of Life in Bangladesh. Am J Trop Med Hyg. 2018 Aug;99(2):489-494. doi: 10.4269/ajtmh.17-0985. Epub 2018 Jun 7. PMID 29893201
- [Background] Faubion WA, Camilleri M, Murray JA, Kelly P, Amadi B, Kosek MN, Enders F, Larson J, Grover M, Boe G, Dyer R, Singh R. Improving the detection of environmental enteric dysfunction: a lactulose, rhamnose assay of intestinal permeability in children aged under 5 years exposed to poor sanitation and hygiene. BMJ Glob Health. 2016 Jul 4;1(1):e000066. doi: 10.1136/bmjgh-2016-000066. eCollection 2016. PMID 28588929
- [Background] Ghosh S, Suri D, Uauy R. Assessment of protein adequacy in developing countries: quality matters. Br J Nutr. 2012 Aug;108 Suppl 2:S77-87. doi: 10.1017/S0007114512002577. PMID 23107551
- [Background] Gibson RS, Ferguson EL, Lehrfeld J. Complementary foods for infant feeding in developing countries: their nutrient adequacy and improvement. Eur J Clin Nutr. 1998 Oct;52(10):764-70. doi: 10.1038/sj.ejcn.1600645. PMID 9805226
- [Background] Goron A, Moinard C. Amino acids and sport: a true love story? Amino Acids. 2018 Aug;50(8):969-980. doi: 10.1007/s00726-018-2591-x. Epub 2018 May 31. PMID 29855718
- [Background] Goto K, Chew F, Torun B, Peerson JM, Brown KH. Epidemiology of altered intestinal permeability to lactulose and mannitol in Guatemalan infants. J Pediatr Gastroenterol Nutr. 1999 Mar;28(3):282-90. doi: 10.1097/00005176-199903000-00013. PMID 10067729
- [Background] Holecek M. Side effects of amino acid supplements. Physiol Res. 2022 Mar 25;71(1):29-45. doi: 10.33549/physiolres.934790. Epub 2022 Jan 19. PMID 35043647
- [Background] Koletzko B, Sauerwald T, Demmelmair H. Safety of stable isotope use. Eur J Pediatr. 1997 Aug;156 Suppl 1:S12-7. doi: 10.1007/pl00014267. PMID 9266209
- [Background] Kosek M, Haque R, Lima A, Babji S, Shrestha S, Qureshi S, Amidou S, Mduma E, Lee G, Yori PP, Guerrant RL, Bhutta Z, Mason C, Kang G, Kabir M, Amour C, Bessong P, Turab A, Seidman J, Olortegui MP, Quetz J, Lang D, Gratz J, Miller M, Gottlieb M. Fecal markers of intestinal inflammation and permeability associated with the subsequent acquisition of linear growth deficits in infants. Am J Trop Med Hyg. 2013 Feb;88(2):390-396. doi: 10.4269/ajtmh.2012.12-0549. Epub 2012 Nov 26. PMID 23185075
- [Background] Kosek MN, Mduma E, Kosek PS, Lee GO, Svensen E, Pan WKY, Olortegui MP, Bream JH, Patil C, Asayag CR, Sanchez GM, Caulfield LE, Gratz J, Yori PP. Plasma Tryptophan and the Kynurenine-Tryptophan Ratio are Associated with the Acquisition of Statural Growth Deficits and Oral Vaccine Underperformance in Populations with Environmental Enteropathy. Am J Trop Med Hyg. 2016 Oct 5;95(4):928-937. doi: 10.4269/ajtmh.16-0037. Epub 2016 Aug 8. PMID 27503512
- [Background] Lee G, Pan W, Penataro Yori P, Paredes Olortegui M, Tilley D, Gregory M, Oberhelman R, Burga R, Chavez CB, Kosek M. Symptomatic and asymptomatic Campylobacter infections associated with reduced growth in Peruvian children. PLoS Negl Trop Dis. 2013;7(1):e2036. doi: 10.1371/journal.pntd.0002036. Epub 2013 Jan 31. PMID 23383356
- [Background] Lee G, Paredes Olortegui M, Penataro Yori P, Black RE, Caulfield L, Banda Chavez C, Hall E, Pan WK, Meza R, Kosek M. Effects of Shigella-, Campylobacter- and ETEC-associated diarrhea on childhood growth. Pediatr Infect Dis J. 2014 Oct;33(10):1004-9. doi: 10.1097/INF.0000000000000351. PMID 25361185
- [Background] Lee GO, McCormick BJJ, Seidman JC, Kosek MN, Haque R, Olortegui MP, Lima AAM, Bhutta ZA, Kang G, Samie A, Amour C, Mason CJ, Ahmed T, Yori PP, Oliveira DB, Alam D, Babji S, Bessong P, Mduma E, Shrestha SK, Ambikapathi R, Lang DR, Gottlieb M, Guerrant RL, Caulfield LE, For The Mal-Ed Network Investigators. Infant Nutritional Status, Feeding Practices, Enteropathogen Exposure, Socioeconomic Status, and Illness Are Associated with Gut Barrier Function As Assessed by the Lactulose Mannitol Test in the MAL-ED Birth Cohort. Am J Trop Med Hyg. 2017 Jul;97(1):281-290. doi: 10.4269/ajtmh.16-0830. PMID 28719336
- [Background] Leenders EKSM, de Waard M, van Goudoever JB. Low- versus High-Dose and Early versus Late Parenteral Amino-Acid Administration in Very-Low-Birth-Weight Infants: A Systematic Review and Meta-Analysis. Neonatology. 2018;113(3):187-205. doi: 10.1159/000481192. Epub 2017 Dec 22. PMID 29268262
- [Background] Lima AA, Brito LF, Ribeiro HB, Martins MC, Lustosa AP, Rocha EM, Lima NL, Monte CM, Guerrant RL. Intestinal barrier function and weight gain in malnourished children taking glutamine supplemented enteral formula. J Pediatr Gastroenterol Nutr. 2005 Jan;40(1):28-35. doi: 10.1097/00005176-200501000-00006. PMID 15625423
- [Background] Louis-Auguste J, Besa E, Zyambo K, Munkombwe D, Banda R, Banda T, Watson A, Mayneris-Perxachs J, Swann J, Kelly P. Tryptophan, glutamine, leucine, and micronutrient supplementation improves environmental enteropathy in Zambian adults: a randomized controlled trial. Am J Clin Nutr. 2019 Nov 1;110(5):1240-1252. doi: 10.1093/ajcn/nqz189. PMID 31504110
- [Background] Marles RJ, Barrett ML, Barnes J, Chavez ML, Gardiner P, Ko R, Mahady GB, Low Dog T, Sarma ND, Giancaspro GI, Sharaf M, Griffiths J. United States pharmacopeia safety evaluation of spirulina. Crit Rev Food Sci Nutr. 2011 Aug;51(7):593-604. doi: 10.1080/10408391003721719. PMID 21793723
- [Background] Martorell R, Khan LK, Schroeder DG. Reversibility of stunting: epidemiological findings in children from developing countries. Eur J Clin Nutr. 1994 Feb;48 Suppl 1:S45-57. PMID 8005090
- [Background] Mbuya MN, Humphrey JH. Preventing environmental enteric dysfunction through improved water, sanitation and hygiene: an opportunity for stunting reduction in developing countries. Matern Child Nutr. 2016 May;12 Suppl 1(Suppl 1):106-20. doi: 10.1111/mcn.12220. Epub 2015 Nov 6. PMID 26542185
- [Background] McCormick BJJ, Murray-Kolb LE, Lee GO, Schulze KJ, Ross AC, Bauck A, Lima AAM, Maciel BLL, Kosek MN, Seidman JC, Ambikapathi R, Bose A, John S, Kang G, Turab A, Mduma E, Bessong P, Shrestra SK, Ahmed T, Mahfuz M, Olortegui MP, Bhutta Z, Caulfield LE; MAL-ED Network Investigators. Intestinal permeability and inflammation mediate the association between nutrient density of complementary foods and biochemical measures of micronutrient status in young children: results from the MAL-ED study. Am J Clin Nutr. 2019 Oct 1;110(4):1015-1025. doi: 10.1093/ajcn/nqz151. PMID 31565748
- [Background] McDonald CM, Manji KP, Gosselin K, Tran H, Liu E, Kisenge R, Aboud S, Fawzi WW, Gewirtz AT, Duggan CP. Elevations in serum anti-flagellin and anti-LPS Igs are related to growth faltering in young Tanzanian children. Am J Clin Nutr. 2016 Jun;103(6):1548-54. doi: 10.3945/ajcn.116.131409. Epub 2016 Apr 27. PMID 27121948
- [Background] McKay S, Gaudier E, Campbell DI, Prentice AM, Albers R. Environmental enteropathy: new targets for nutritional interventions. Int Health. 2010 Sep;2(3):172-80. doi: 10.1016/j.inhe.2010.07.006. PMID 24037697
- [Background] Millward DJ, Layman DK, Tome D, Schaafsma G. Protein quality assessment: impact of expanding understanding of protein and amino acid needs for optimal health. Am J Clin Nutr. 2008 May;87(5):1576S-1581S. doi: 10.1093/ajcn/87.5.1576S. PMID 18469291
- [Background] Owino V, Ahmed T, Freemark M, Kelly P, Loy A, Manary M, Loechl C. Environmental Enteric Dysfunction and Growth Failure/Stunting in Global Child Health. Pediatrics. 2016 Dec;138(6):e20160641. doi: 10.1542/peds.2016-0641. Epub 2016 Nov 4. PMID 27940670
- [Background] Philpott H, Nandurkar S, Lubel J, Gibson PR. Alternative investigations for irritable bowel syndrome. J Gastroenterol Hepatol. 2013 Jan;28(1):73-7. doi: 10.1111/j.1440-1746.2012.07291.x. PMID 23033865
- [Background] Platts-Mills JA, Babji S, Bodhidatta L, Gratz J, Haque R, Havt A, McCormick BJ, McGrath M, Olortegui MP, Samie A, Shakoor S, Mondal D, Lima IF, Hariraju D, Rayamajhi BB, Qureshi S, Kabir F, Yori PP, Mufamadi B, Amour C, Carreon JD, Richard SA, Lang D, Bessong P, Mduma E, Ahmed T, Lima AA, Mason CJ, Zaidi AK, Bhutta ZA, Kosek M, Guerrant RL, Gottlieb M, Miller M, Kang G, Houpt ER; MAL-ED Network Investigators. Pathogen-specific burdens of community diarrhoea in developing countries: a multisite birth cohort study (MAL-ED). Lancet Glob Health. 2015 Sep;3(9):e564-75. doi: 10.1016/S2214-109X(15)00151-5. Epub 2015 Jul 19. PMID 26202075
- [Background] Prendergast AJ, Humphrey JH. The stunting syndrome in developing countries. Paediatr Int Child Health. 2014 Nov;34(4):250-65. doi: 10.1179/2046905514Y.0000000158. Epub 2014 Oct 13. PMID 25310000
- [Background] Prentice AM, Ward KA, Goldberg GR, Jarjou LM, Moore SE, Fulford AJ, Prentice A. Critical windows for nutritional interventions against stunting. Am J Clin Nutr. 2013 May;97(5):911-8. doi: 10.3945/ajcn.112.052332. Epub 2013 Apr 3. PMID 23553163
- [Background] Psaki SR, Seidman JC, Miller M, Gottlieb M, Bhutta ZA, Ahmed T, Ahmed AS, Bessong P, John SM, Kang G, Kosek M, Lima A, Shrestha P, Svensen E, Checkley W; MAL-ED Network Investigators. Measuring socioeconomic status in multicountry studies: results from the eight-country MAL-ED study. Popul Health Metr. 2014 Mar 21;12(1):8. doi: 10.1186/1478-7954-12-8. PMID 24656134
- [Background] Regassa R, Tamiru D, Duguma M, Belachew T. Environmental enteropathy and its association with water sanitation and hygiene in slum areas of Jimma Town Ethiopia. PLoS One. 2023 Jun 23;18(6):e0286866. doi: 10.1371/journal.pone.0286866. eCollection 2023. PMID 37352168
- [Background] Richard SA, McCormick BJJ, Murray-Kolb LE, Lee GO, Seidman JC, Mahfuz M, Ahmed T, Guerrant RL, Petri WA, Rogawski ET, Houpt E, Kang G, Mduma E, Kosek MN, Lima AAM, Shrestha SK, Chandyo RK, Bhutta Z, Bessong P, Caulfield LE; MAL-ED Network Investigators. Enteric dysfunction and other factors associated with attained size at 5 years: MAL-ED birth cohort study findings. Am J Clin Nutr. 2019 Jul 1;110(1):131-138. doi: 10.1093/ajcn/nqz004. PMID 31127812
- [Background] Rom O, Liu Y, Liu Z, Zhao Y, Wu J, Ghrayeb A, Villacorta L, Fan Y, Chang L, Wang L, Liu C, Yang D, Song J, Rech JC, Guo Y, Wang H, Zhao G, Liang W, Koike Y, Lu H, Koike T, Hayek T, Pennathur S, Xi C, Wen B, Sun D, Garcia-Barrio MT, Aviram M, Gottlieb E, Mor I, Liu W, Zhang J, Chen YE. Glycine-based treatment ameliorates NAFLD by modulating fatty acid oxidation, glutathione synthesis, and the gut microbiome. Sci Transl Med. 2020 Dec 2;12(572):eaaz2841. doi: 10.1126/scitranslmed.aaz2841. PMID 33268508
- [Background] Ryan KN, Stephenson KB, Trehan I, Shulman RJ, Thakwalakwa C, Murray E, Maleta K, Manary MJ. Zinc or albendazole attenuates the progression of environmental enteropathy: a randomized controlled trial. Clin Gastroenterol Hepatol. 2014 Sep;12(9):1507-13.e1. doi: 10.1016/j.cgh.2014.01.024. Epub 2014 Jan 22. PMID 24462483
- [Background] Sangalang SO, Lemence ALG, Ottong ZJ, Valencia JC, Olaguera M, Canja RJF, Mariano SMF, Prado NO, Ocana RMZ, Singson PAA, Cumagun ML, Liao J, Anglo MVJC, Borgemeister C, Kistemann T. School water, sanitation, and hygiene (WaSH) intervention to improve malnutrition, dehydration, health literacy, and handwashing: a cluster-randomised controlled trial in Metro Manila, Philippines. BMC Public Health. 2022 Nov 7;22(1):2034. doi: 10.1186/s12889-022-14398-w. PMID 36344973
- [Background] Lee GO, Schillinger R, Shivakumar N, Whyte S, Huq S, Ochieng Konyole S, Chileshe J, Paredes-Olortegui M, Owino V, Yazbeck R, Kosek MN, Kelly P, Morrison D. Optimisation, validation and field applicability of a 13C-sucrose breath test to assess intestinal function in environmental enteropathy among children in resource poor settings: study protocol for a prospective study in Bangladesh, India, Kenya, Jamaica, Peru and Zambia. BMJ Open. 2020 Nov 17;10(11):e035841. doi: 10.1136/bmjopen-2019-035841. PMID 33203623
- [Background] Shivakumar N, Kashyap S, Jahoor F, Devi S, Preston T, Thomas T, Kurpad AV. The Systemic Availability of Indispensable Amino Acids from Orally Ingested Algal and Legume Protein in Young Children at Risk of Environmental Enteric Dysfunction. Am J Clin Nutr. 2023 Jul;118(1):96-102. doi: 10.1016/j.ajcnut.2023.05.014. Epub 2023 May 11. PMID 37178715
- [Background] Shivakumar N, Thomas T, Devi S, Jahoor F, Kurpad AV. Free living total energy expenditure in young South Indian children at risk of environmental enteric dysfunction and its relation to faltered linear growth. Eur J Clin Nutr. 2023 May;77(5):532-537. doi: 10.1038/s41430-023-01268-w. Epub 2023 Jan 31. PMID 36720933
- [Background] Smith HE, Ryan KN, Stephenson KB, Westcott C, Thakwalakwa C, Maleta K, Cheng JY, Brenna JT, Shulman RJ, Trehan I, Manary MJ. Multiple micronutrient supplementation transiently ameliorates environmental enteropathy in Malawian children aged 12-35 months in a randomized controlled clinical trial. J Nutr. 2014 Dec;144(12):2059-65. doi: 10.3945/jn.114.201673. Epub 2014 Oct 1. PMID 25411039
- [Background] Smriga M. International Regulations on Amino Acid Use in Foods and Supplements and Recommendations to Control Their Safety Based on Purity and Quality. J Nutr. 2020 Oct 1;150(Suppl 1):2602S-2605S. doi: 10.1093/jn/nxaa093. PMID 33000158
- [Background] Terry R, van Wettere WH, Whittaker AL, Herde PJ, Howarth GS. Using the noninvasive (13)C-sucrose breath test to measure intestinal sucrase activity in swine. Comp Med. 2012 Dec;62(6):504-7. PMID 23561884
- [Background] Trehan I, Kelly P, Shaikh N, Manary MJ. New insights into environmental enteric dysfunction. Arch Dis Child. 2016 Aug;101(8):741-4. doi: 10.1136/archdischild-2015-309534. Epub 2016 Mar 1. PMID 26933151
- [Background] Joint WHO/FAO/UNU Expert Consultation. Protein and amino acid requirements in human nutrition. World Health Organ Tech Rep Ser. 2007;(935):1-265, back cover. PMID 18330140